CLINICAL TRIAL: NCT01750619
Title: Clinical Outcomes of the Endoscopic Resection of Premalignant and Malignant Gastrointestinal Lesions
Status: Recruiting | Type: Observational
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Kenneth Binmoeller, Interventional Endoscopy Services Program Director, California Pacific Medical Center Research Institute
Other Study IDs: 2011.090
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Gastrointestinal Neoplasms; Benign Neoplasm of Intestinal Tract
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mucosal tumors of the colon: Patients who received endoscopic treatment for noninvasive mucosal tumors of the colon.
- Nonampullary tumors of the duodenum: Patients who received endoscopic treatment for noninvasive mucosal tumors of the duodenum.
- Ampullary tumors: Patients who received endoscopic treatment for noninvasive ampullary tumors.

SUMMARY:
To evaluate clinical outcome for patients receiving treatment of suspected premalignant and malignant gastrointestinal lesions at Interventional Endoscopy Services. The primary outcome is curative endoscopic resection. Secondary outcomes include resection technique utilized, rates of en bloc resection and adverse event rates, including infection, bleeding, perforation and death, and one-year survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years that have been referred for endoscopic treatment of GI lesions.

Exclusion Criteria:

* Patients for whom endoscopic treatment was not performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Interventional Endoscopy Services at CPMC for treatment of GI tract tumors.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-07; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Technical success. | 1 day to 3 months
  Technical success is defined as complete resection confirmed by the endoscopic absence of adenomatous tissue after inspection with high-definition white light and narrow-band imaging.

SECONDARY OUTCOMES:
Short term recurrence rate | Less than 1 year
  Freedom from recurrence on follow-up endoscopy with high definition white light and narrow band imaging and on mucosal biopsies of the endoscopic mucosal resection site
Long term recurrence rate | Greater than 1 year
  Freedom from recurrence on follow-up endoscopy with high definition white light and narrow band imaging and on mucosal biopsies of the endoscopic mucosal resection site
Adverse event rate | up to 1 month post procedure.
  Adverse events include infection, bleeding, perforation and death.
Endoscopic en bloc resection rate | Immediate
  Resection in 1 piece without fragmentation, along or extrinsic to the diathermic markings placed around the perimeter of the lesion before resection, without remnant abnormal tissue visible on HD white-light imaging or NBI

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth F Binmoeller, M.D., Principal Investigator — California Pacific Medical Center
Locations (1):
- Interventional Endoscopy Services, San Francisco, California, United States

REFERENCES:
- [Derived] Binmoeller KF, Hamerski CM, Shah JN, Bhat YM, Kane SD. Underwater EMR of adenomas of the appendiceal orifice (with video). Gastrointest Endosc. 2016 Mar;83(3):638-42. doi: 10.1016/j.gie.2015.08.079. Epub 2015 Sep 14. PMID 26375437
- [Derived] Binmoeller KF, Hamerski CM, Shah JN, Bhat YM, Kane SD, Garcia-Kennedy R. Attempted underwater en bloc resection for large (2-4 cm) colorectal laterally spreading tumors (with video). Gastrointest Endosc. 2015 Mar;81(3):713-8. doi: 10.1016/j.gie.2014.10.044. PMID 25708759